CLINICAL TRIAL: NCT03593876
Title: Strategy Training for People With Aphasia After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Given the design of the study, we reached saturation with a sample of 16
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Skidmore, PhD, OTR/L, Professor and Chair, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO18050075; R01HD074693 (NIH)
Record Dates: First submitted 2018-06-22; First posted 2018-07-20 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Strategy Training
Keywords: Stroke; Aphasia; Rehabilitation; Cognition; Disability
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strategy Training (Experimental): Strategy training is a form of meta-cognitive instruction that trains individuals with stroke-related cognitive impairments to identify and prioritize problematic daily activities, identify the barriers impeding performance, generate and evaluate their own strategies to address barriers, and apply these skills through iterative practice.
  Interventions: Behavioral: Strategy Training

INTERVENTIONS:
Behavioral: Strategy Training — This study will use an adapted form of strategy training for people with communication impairments.

SUMMARY:
One-third to one-half of acute strokes result in newly acquired cognitive impairments. Approximately 30 to 40% of people in the acute phase of stroke also sustain communication impairments. Stroke-related cognitive impairments are associated with significant functional disability, as indicated by the inability to regain independence in daily activities. The overall aim of this study is to examine the feasibility of an adapted form of strategy training for people with communication impairments who are admitted to inpatient rehabilitation. These analyses will address a critical gap in current rehabilitation research, namely the exclusion of people with communication impairments in acute stroke rehabilitation clinical trials, and provide pilot data to inform the design of future inclusive clinical trials seeking to reduce disability after stroke.

DETAILED DESCRIPTION:
This pilot study will use a descriptive case series design with repeated measures to assess the feasibility of an adapted form of strategy training for people with communication impairments after acute stroke. The investigators will recruit people with aphasia due to stroke admitted to the inpatient rehabilitation units and administer the adapted form of strategy training one session per day 5 days per week for 10-15 sessions. The investigators will assess the feasibility of the intervention based on feedback from participants and therapists. These data will serve as pilot data to inform the design of a future clinical trials for people with cognitive impairments after stroke, including people with communication impairments. These efforts will allow the investigators to test new models to support optimal interventions for individuals with stroke-related cognitive impairments, including people with communication impairments who are among those most vulnerable for long-term disability.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of acute stroke
* admission to acute rehabilitation
* mild to moderate aphasia but able to understand and express communication with verbal, written, and/or augmentative communication (score of 1 or 2 on the National Institutes of Health Stroke Scale item 9, or score 1 to 5 on the Boston Diagnostic Aphasia Examination Severity Scale)

Exclusion Criteria:

* pre-stroke diagnosis of dementia
* severe global aphasia (Boston Diagnostic Aphasia Examination Severity Scale score of 0)
* dysarthria as the only communication impairment (score of 1 or 2 two on the National Institutes of Health Stroke Scale item 10, but score of 0 on item 9)
* current major depressive disorder (unless treated and in partial remission), bipolar disorder, or any other psychotic disorder (indicated by PRIME-MD)severe global aphasia (Boston Diagnostic Aphasia Examination Severity Scale score of 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R. Skidmore, PhD, OTR/L, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Strategy Training: Strategy training is a form of meta-cognitive instruction that trains individuals with stroke-related cognitive impairments to identify and prioritize problematic daily activities, identify the barriers impeding performance, generate and evaluate their own strategies to address barriers, and apply these skills through iterative practice.
  Strategy Training: This study will use an adapted form of strategy training for people with communication impairments. Supported conversation principles will be standardized and incorporated into the intervention protocol.
Period: Overall Study
Arm/Group | Strategy Training
Started | 16
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Discharged home before intervention completion | 2

BASELINE CHARACTERISTICS:
Arm/Group | Strategy Training
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Comorbidity, Charlson Comorbidity Index [Mean (Standard Deviation); unit: total score] — Comordity severity (measured with the Charlson Comorbidity Index) assesses the presence of 21 comorbid conditions using a scale of 0 (absent) to 1 (present) for each condition. Total scores range from 0 to 21. Higher values represent more severe comorbidity.
  total score | 2.3 (1.7)
Chronicity, Days since stroke [Mean (Standard Deviation); unit: days] | 25.6 (27.6)
Stroke Hemisphere, Left [Number; unit: participants] | 13
Inpatient Rehabilitation Length of Stay, Days [Mean (Standard Deviation); unit: days] | 22.5 (9.6)
Aphasia Severity, Boston Diagnostic Aphasia Examination Severity Scale [Mean (Standard Deviation); unit: total score] — Aphasia severity (measured with the Boston Diagnostic Aphasia Examination Severity Scale) is assessed using a single scale of 0 (no usable speech or auditory comprehension) to 5 (minimal discernible speech impairments; subjective difficulties not apparent to listener). Higher values represent lower aphasia severity.
  total score | 1.9 (1.1)
Stroke Severity, National Institutes of Health Stroke Scale [Mean (Standard Deviation); unit: total score] — Stroke severity (measured with the National Institutes of Health Stroke Scale) is assessed through 15 items addressing a range of neurological impairments that emerge after stroke (cognition, motor function, sensory function, language, perception). The total score ranges from 0 (no neurological impairment) to 42 (severe neurological impairment). Higher values represent greater stroke severity.
  total score | 8.6 (5.2)
Disability, Functional Independence Measure [Mean (Standard Deviation); unit: total score] — Disability (measured with the Functional Independence Measure) is assessed through 18 tasks in 6 functional domains (self-care, sphincter control, transfers, locomotion, communication and social cognition) using a scale of 1 (dependent) to 7 (independent). Scores range from 18 to 126. Higher values represent better outcomes.
  total score | 52.4 (21.0)
Cognitive Linguistic Quick Test Executive Function Score [Mean (Standard Deviation); unit: composite score] — Cognition (measured with the Cognitive Linguistic Quick Test Executive Function Score) is measured with 4 tasks (symbol trails, generative naming, mazes, and design generation). The severity score ranges from 40 (within normal limits) to 0 (severe impairment). Higher values represent better outcomes.
  composite score | 12.6 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Patient-therapist Communication Score
Description: Measure of Participation in Conversation (MPC) Interaction score greater than or equal to 2. The scale assesses the degree of participation executed by the participant with communication impairment during supported conversation. Scores range from 0=no participation/comprehension to 4=full participation/comprehension.
Time Frame: Baseline to Post-Intervention (up to 3 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strategy Training
Number analyzed (Participants) | 13
score on a scale | 3.0 (1.0)
Statistical Analysis 1: Comparison: Strategy Training; Test type: Other; The a priori analysis plan was to defer statistical or hypothesis testing due to the focus on feasibility, and rather to assess mean participant-therapist communication scores across intervention sessions. The mean and standard deviation of these scores was 3.00 (1.00). The a priori criterion for feasibility was a mean score of 2.0 or greater

2. Secondary Outcome: Change in Independence With Daily Activities
Description: Change in independence measured with the Functional Independence Measure. The FIM assesses 18 tasks in 6 functional domains (self-care, sphincter control, transfers, locomotion, communication and social cognition) using a scale of 1 (dependent) to 7 (independent). Scores range from 18 to 126. Higher values represent better outcomes. The a priori criterion for change was a medium effect size of change (Cohen's d≥0.5).
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Strategy Training
Number analyzed (Participants) | 13
change score on a scale | 51.7 (21.0)
Statistical Analysis 1: Comparison: Strategy Training; The a priori analysis plan was to defer statistical or hypothesis testing due to the focus on feasibility, and rather to assess change scores and effect size of the change scores to compare with previously published clinical trials; Test type: Other; Mean Difference (Net) = 51.71, Standard Deviation 21.04; The repeated measures effect size of change was Cohen's d(rm)=3.08

3. Secondary Outcome: Change in Cognition
Description: Change in cognition measured with the Cognitive Linguistic Quick Test Executive Function Score. The severity score measures executive functions using 4 tasks (symbol trails, generative naming, mazes, and design generation). The score ranges from 40 (within normal limits) to 0 (severe impairment). Higher values represent better outcomes. The a priori criterion for change was a medium effect size of change (Cohen's d≥0.5).
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: composite score
Arm/Group | Strategy Training
Number analyzed (Participants) | 13
composite score | 1.8 (3.5)
Statistical Analysis 1: Comparison: Strategy Training; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mean Difference (Net) = 11.02, Standard Deviation 7.24; The repeated measures effect size of change, Cohen's d(rm)=1.70

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Strategy Training
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03593876/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03593876/SAP_001.pdf
  • Informed Consent Form (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03593876/ICF_002.pdf